CLINICAL TRIAL: NCT00486850
Title: Synchronized Intermittent Mandatory Ventilation (SIMV) Versus Nasal Intermittent Positive Pressure Ventilation (NIPPV) In Preterm Infants With Respiratory Distress
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Dey, L.P., Napa Valley, Califonia (Unknown)
Responsible Party: Rangasamy Ramanathan, MD., University of Southern California
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIMV versus NIPPV Trial
Record Dates: First submitted 2007-06-13; First posted 2007-06-15 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-02

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: RDS; Preterm; SIMV; NIPPV
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Extubation to Nasal IPPV — Comparison of extubation to NIPPV versus NCPAP
  Other Names: NIPPV; SIMV

SUMMARY:
Title of Study: A Prospective, Randomized, Multicenter Trial Comparing Synchronized Intermittent Mandatory Ventilation (SIMV) vs. Early Extubation to Nasal Intermittent Positive Pressure Ventilation (NIPPV) after Surfactant Treatment in Preterm Infants with Respiratory Distress Treatment Period (Planned): 7 days Objectives: To compare the impact of early extubation [within 120 minutes of birth to Nasal Intermittent Positive Pressure Ventilation (NIPPV group) vs. Synchronized Intermittent Mandatory Ventilation (SIMV group) on the incidence of mechanical ventilation via endotracheal tube at 7 days of age in 26 to 29 + 6 weeks gestation premature infants with respiratory distress treated with intratracheal Curosurf (poractant alpha) within 60 minutes of birth.

Secondary objectives include evaluation of overall clinical outcomes at 7 days, 28 days, and 36 weeks postmenstrual age (PMA) and/or at discharge, complications, safety, and adverse events.

Number of Subjects: 110

DETAILED DESCRIPTION:
Respiratory management: SIMV group:

Infants randomized to SIMV will be maintained on SIMV per standard unit protocol. Infant can be progressively weaned and extubated to NCPAP if infant meets the minimum criteria for extubation. Caffeine will be administered around the time of extubation.

NIPPV group:

Extubated to NIPPV within 120 minutes of birth if the fraction of inspired oxygen (FiO2) is less than 0.60 after the first dose of surfactant. Caffeine will be administered around the time of extubation. Infant can be reintubated if clinical parameters necessitate mechanical ventilation. NIPPV may be discontinued when patients are weaned to a positive end expiratory pressure of 5 cmsH20 with back up rate <10 bpm and FiO2 <0.30 for 24 hours to nasal continuous positive airway pressure (NCPAP).

Surfactant administration:

Prior to randomization and enrollment, infants will receive an initial dose of poractant alfa 200mg/kg. Subsequent doses of 100mg/kg can be given 12 hours after the initial dose based upon clinical criteria. Up to 2 additional doses can be given within 48 hours of age in infants who remain intubated.

Criteria for Evaluation Primary Endpoint: The need for mechanical ventilation via the endotracheal tube at 7 days of age.

Secondary Endpoints: Additional doses of surfactant, duration (days) of mechanical ventilation, duration (days) of supplemental oxygen, days on NIPPV, days on CPAP, use of postnatal steroids for bronchopulmonary dysplasia (BPD), death before discharge, pneumothorax, pneumomediastinum, pneumopericardium, pulmonary hemorrhage, patent ductus arteriosis (PDA), intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), growth (weight on day 28 and 36 weeks PMA, and/or discharge), length of hospital stay.

Adverse events (AEs) and serious adverse events (SAEs) will be monitored, collected, analyzed, and reported.

Safety will be monitored throughout the study and will be based on prospectively defined complications (safety outcomes) and will allow for reporting of as yet unidentified potential complications.

All AEs and SAEs will be reported, with SAEs reported on an expedited basis per regulatory requirements and timeframes to the responsible investigational review boards (IRBs), and the Data Safety Monitoring Board (DSMB). Interim analysis will be performed by an independent statistician after 50 patients are enrolled and data will be submitted to the DSMB members. They will monitor for any adverse events, specifically, mortality and make a recommendation about continuation of the study. The DSMB will not disclose any findings to avoid any biases except to issuing a continue or discontinue statement. If there is a statistically significant difference in the primary endpoint- the need for mechanical ventilation via endotracheal tube at 7 days of age (p < 0.02) or statistically higher incidence in mortality within one of the treatment groups, the trial can be closed and these midpoint results will be disclosed.

Statistical Methods Sample Size: A sample size of 100 patients is needed. The need for mechanical ventilation via endotracheal tube at 7 days of age in this preterm population has been reported to range between 63% (Verder 1999) and 43% (Dani 2004). On the basis of data collected from our own center and from published data in VLBW infants, a sample size of 50 infants in each group will be needed to demonstrate a 50% reduction in the need for mechanical ventilation via endotracheal tube at 7 days of age (power of 0.8 and an α-error of 0.05). An additional 10 patients (10%) will be allowed for to accommodate for dropouts.

Primary Endpoint: Analyses of the primary endpoint will be based on intention to treat (ITT) analysis of all randomized, eligible subjects. Statistical analyses will be performed by using Student's t test for continuous normally distributed variables and with the Wilcoxon rank sum test for non-parametric variables. Comparison of proportions and analysis of categorical variables will be performed using 2-tailed Fisher's exact test and logistic regression analysis. A p value of < 0.05 will be considered statistically significant.

Secondary Endpoints: The secondary efficacy analyses will be performed using the ITT population. The following secondary variables that will be analyzed include need for additional doses of surfactant, duration of mechanical ventilation and supplemental oxygen, days on nasal CPAP, postnatal steroid use for BPD, growth (weight on day 28 and 36 weeks PMA, and/or discharge) and length of hospital stay. A p-value of less than 0.05 will be considered significant for testing the effect of each factor. A multiple regression analysis may be employed as required if confounding effects are identified within the study (e.g., gestational age, race, center, antenatal or postnatal steroid use).

ELIGIBILITY:
Inclusion Criteria:

1. Estimated gestational age 26 to 29 + 6 weeks inclusive;
2. Inborn;
3. Birth Weight: ≥ 600 grams;
4. Required endotracheal intubation for respiratory distress;
5. Has received one dose of poractant alfa 200mg/kg within 60 minutes of birth;
6. No known lethal congenital anomaly or genetic syndromes;
7. No known lung maturity; and
8. Signed parental informed consent

Exclusion Criteria:

1. Gestational age < 26 weeks or ≥ 30 weeks;
2. Birth weight less than 600 grams;
3. Apgar score of 0 at one minute of age; and
4. Lethal congenital anomaly or genetic syndrome identified antenatally or within 60 minutes of birth

Ages: 10 Minutes to 120 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2006-10; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Mechanical Ventilation via endotracheal tube at 7 days of age | At 7 days of age

SECONDARY OUTCOMES:
Overall clinical outcomes at 7 days, 28 days, and 36 weeks postmenstrual age | At 7 days, 28 days and at 36 weeks postmenstraul age

CONTACTS AND LOCATIONS:
Overall Officials: Rangasamy Ramanathan, MD, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - Women's and Children's Hospital, Room l-919, 1240, N.Mission Road, Los Angeles, California
  - Sharp Mary Birch Hospital for Women, San Diego, California
  - Medical College of Georgia, Augusta, Georgia
  - Children's Hospital, OUMC, Oklahoma City, Oklahoma